CLINICAL TRIAL: NCT05198934
Title: A Phase 3 Multicenter, Randomized, Open-label, Active-controlled Study of Sotorasib and Panitumumab Versus Investigator's Choice (Trifluridine and Tipiracil, or Regorafenib) for the Treatment of Previously Treated Metastatic Colorectal Cancer Subjects With Kirsten Rat Sarcoma (KRAS) p.G12C Mutation
Brief Title: Sotorasib and Panitumumab Versus Investigator's Choice for Participants With Kirsten Rat Sarcoma (KRAS) p.G12C Mutation
Acronym: CodeBreak300
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190172; 2024-511187-81-00 (EU CTIS Number)
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Sotorasib; AMG 510; Panitumumab; Metastatic colorectal cancer; Kirsten rat sarcoma p.G12C mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sotorasib; Panitumumab; trifluridine tipiracil drug combination; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Sotorasib 960 mg QD + panitumumab (Experimental)
  Interventions: Drug: Sotorasib; Drug: Panitumumab
- Arm B: Sotorasib 240 mg QD + panitumumab (Experimental)
  Interventions: Drug: Sotorasib; Drug: Panitumumab
- Arm C : Investigator's choice (Active Comparator): Participants will be administered trifluridine and tipiracil, or regorafenib
  Interventions: Drug: Trifluridine and Tipiracil; Drug: Regorafenib

INTERVENTIONS:
Drug: Sotorasib — Sotorasib will be administered orally
  Other Names: AMG 510, Lumakras, Lumykras
  Arms: Arm A: Sotorasib 960 mg QD + panitumumab; Arm B: Sotorasib 240 mg QD + panitumumab
Drug: Panitumumab — Panitumumab will be administered as intravenous (IV) infusion
  Other Names: Vectibix
  Arms: Arm A: Sotorasib 960 mg QD + panitumumab; Arm B: Sotorasib 240 mg QD + panitumumab
Drug: Trifluridine and Tipiracil — Trifluridine and Tipiracil will be administered orally
  Other Names: Lonsurf
  Arms: Arm C : Investigator's choice
Drug: Regorafenib — Regorafenib will be administered orally
  Other Names: Stivarga
  Arms: Arm C : Investigator's choice

SUMMARY:
The aim of the study is to compare progression-free survival (PFS) in previously treated participants with Kirsten rat sarcoma (KRAS) p.G12C mutated colorectal cancer (CRC) receiving sotorasib 240 mg once daily (QD) and panitumumab vs investigator's choice (trifluridine and tipiracil, or regorafenib), and sotorasib 960 mg QD and panitumumab vs investigator's choice (trifluridine and tipiracil, or regorafenib).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent/assent prior to initiation of any study specific activities/procedures.
* Age ≥18 years.
* Pathologically documented metastatic colorectal adenocarcinoma with Kirsten rat sarcoma (KRAS) p.G12C mutation as determined by prospective central testing, using the analytically validated Qiagen Therascreen KRAS RGQ polymerase chain reaction Kit in CRC as an investigational device demonstrating a KRAS p.G12C mutation is present. Local testing and documentation of KRAS p.G12C mutation should have been previously performed as part of standard of care.
* Participants will have received at least 1 prior line of therapy for metastatic disease. Participants must have received and progressed or experienced disease recurrence on or after fluoropyrimidine, irinotecan, and oxaliplatin given for metastatic disease unless the participant, in the opinion of the investigator, is not a candidate for fluoropyrimidine, irinotecan, or oxaliplatin, in which case, the participant may be eligible after investigator discussion with Amgen medical monitor provided participant has received at least one prior line of therapy for metastatic disease and provided trifluridine and tipiracil or regorafenib is deemed the appropriate next line of therapy for the participant.
* Measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria. Lesions previously radiated are not considered measurable unless they have progressed after radiation.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2.
* Life expectancy of >3 months, in the opinion of the investigator.
* Adequate hematologic and end-organ function, defined as the following within 2 weeks prior to cycle 1 day 1:

  * Absolute neutrophil count (ANC) ≥1.5 x 10^9/L (without granulocyte colony stimulating factor support within 2 weeks of laboratory test used to determine eligibility).
  * Hemoglobin ≥9.0 g/dL (without transfusion within 2 weeks of laboratory test used to determine eligibility).
  * Platelet count ≥100 x 10^9/L (without transfusion within 2 weeks of laboratory test used to determine eligibility).
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal (ULN).
  * Serum bilirubin ≤1.0 x ULN. For participants with Gilbert's disease, total bilirubin or direct bilirubin needs to be ≤1.0 x ULN.
  * International normalized ratio (INR) and activated partial thromboplastin time (or partial thromboplastin time) ≤1.5 x ULN. Prothrombin time (PT) ≤1.5 x ULN may be used instead of INR for sites whose labs do not report INR.
  * Estimated glomerular filtration rate based on Modification of Diet in Renal Disease (MDRD) calculation ≥30 mL/min/1.73 m^2.
* Fridericia's Correction Formula (QTcF) ≤470 msec.

Exclusion Criteria:

* Active brain metastases. Participants who have had brain metastases resected or have received radiation therapy ending at least 4 weeks prior to study day 1 are eligible if they meet all of the following criteria: a) residual neurological symptoms grade ≤2; b) on stable doses of dexamethasone or equivalent for at least 2 weeks, if applicable; and c) follow-up magnetic resonance imaging (MRI) performed within 28 days of day 1 shows no progression or new lesions appearing.
* History or presence of hematological malignancies unless curatively treated with no evidence of disease ≥2 years.
* History of other malignancy within the past 3 years, with the following exceptions:

  * Malignancy treated with curative intent and with no known active disease present for ≥3 years before enrollment and felt to be at low risk for recurrence by the treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
  * Adequately treated breast ductal carcinoma in situ without evidence of disease.
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
  * Adequately treated urothelial papillary non-invasive carcinoma or carcinoma in situ.
* Leptomeningeal disease.
* Significant gastrointestinal (GI) disorder that results in significant malabsorption, requirement for intravenous (IV) alimentation, or inability to take oral medication.
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 6 months prior to randomization, unstable arrhythmias or unstable angina.
* Previous treatment with a KRAS G12C inhibitor.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Approximately 3 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 3 years
Objective Response Rate (ORR) | Approximately 3 years
Duration of Response (DOR) | Approximately 3 years
Time to Response (TTR) | Approximately 3 years
Disease Control Rate (DCR) | Approximately 3 years
Investigator Assessed ORR | Approximately 3 years
Investigator Assessed PFS | Approximately 3 years
Number of Participants with a Treatment-emergent Adverse Event (TEAE) | Approximately 3 years
  A TEAE is any untoward medical occurrence in a clinical study participant following first dose of treatment irrespective of a causal relationship with the study treatment. Any clinically significant changes in vital signs and clinical laboratory tests following first dose will be recorded as TEAEs.
Change from Baseline in Fatigue Severity as Measured by Item 3 of the Brief Fatigue Inventory (BFI) | Baseline and Week 8
  Item 3 of the BFI records a participants' fatigue on a scale from 0 to 10. Higher scores indicate a higher severity of fatigue. An increase in score from baseline indicates a worsening of fatigue. A decrease in score from baseline indicates an improvement in fatigue.
Change from Baseline in Pain Severity as Measured by Item 3 of the Brief Pain Inventory (BPI) | Baseline and Week 8
  Item 3 of the BPI records a participants' pain on a scale from 1 to 10, where pain is mild (score of 1 to 4), moderate (score of 5 to 6), or severe (score of 7 to 10). An increase in score from baseline indicates a worsening of pain. A decrease in score from baseline indicates a lessening of pain.
Change from Baseline in Physical Functioning as Measured by the Physical Function Domain of the European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire-Core Questionnaire (EORTC QLQ-C30) | Baseline and Week 8
  The physical function domain of the EORTC QLQ-C30 assesses a participants' quality of life regarding their physical function on a scale from 1 to 4, with higher scores indicating a worse outcome. An increase in score from baseline indicates a worsening of physical functioning. A decrease in score from baseline indicates an improvement in physical functioning.
Change from Baseline in Global Health Status as Measured by Questions 29 and 30 of the EORTC QLQ-C30 | Baseline and Week 8
  Questions 29 and 30 of the EORTC QLQ-C30 assess a participants' global health status on a scale from 1 to 7, with higher scores indicating a better outcome. An increase in score from baseline indicates an improvement in global health status. A decrease in score from baseline indicates a worsening in global health status.
Change from Baseline For All Subscales of the BFI | Baseline and Week 8
  The BFI is a questionnaire that includes 3 items to assess fatigue severity and 5 items to assess interference due to fatigue, with each item reported on a numeric rating scale from 0 to 10. Higher scores indicate a higher severity of fatigue. An increase in score from baseline indicates a worsening of fatigue. A decrease in score from baseline indicates an improvement in fatigue.
Change from Baseline For All Subscales of the BPI | Baseline and Week 8
  The BPI is a 9-item questionnaire which includes 2 body diagrams, four items to assess pain severity, four items to assess pain interference and one question about percentage of pain relief by analgesics. The level of pain and pain interference assessed can be divided into categories based on score of mild (1 to 4), moderate (5 to 6), and severe (7 to 10). An increase in score from baseline indicates a worsening of pain. A decrease in score from baseline indicates a lessening of pain.
Change from Baseline For All Subscales and Domains of EORTC QLQ-C30 | Baseline and Week 8
  The EORTC QLQ-C30 is a self-reporting 30-item generic instrument which assesses 5 functional domains (physical, role, emotional, cognitive, social), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties), and a global health status/quality of life (QOL) scale. Higher scores indicate a worse outcome. An increase in score from baseline indicates a worsening of outcome. A decrease in score from baseline indicates an improvement in outcome.
Change from Baseline in Visual Analog Scale (VAS) Scores as Measured by EuroQol-5D level 5 (EQ-5D-5L) | Baseline and Week 8
  The EQ-5D-5L questionnaire is a 2-page, standardized instrument for use as a measure of health outcome. It is comprised of a 5-dimension health status measure and a visual analogue scale. The 5-dimension health status measure evaluates: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression based on a 5-level scale: no problems, slight problems, moderate problems, severe problems, and extreme problems. The visual analogue scale records the participant's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
Average Score on Single Question on Symptom Bother GP5 from Functional Assessment of Cancer Therapy - General (FACT-G) | Approximately 2 years
  The GP5 from the FACT-G is a single item included in the Physical Well-Being subscale of the FACT-G. Responses to the item: "I am bothered by side effects of treatment" are rated on a 5-point Likert scale from "not at all" to "very much".
Average Score of Patient Global Impression of Change (PGIC) | Approximately 2 years
  The PGIC scale consists of one item which measures the participants' perception of change in their condition relative to the beginning of the study. Responses are rated on a 7-item response scale ranging from very much improved to very much worse.
Maximum Plasma Concentration (Cmax) of Sotorasib | Day 1 to approximately 2 years
Cmax of Panitumumab | Day 1 to approximately 2 years
Area Under the Plasma Concentration-time Curve (AUC) of Sotorasib | Day 1 to approximately 2 years
AUC of Panitumumab | Day 1 to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (105):
- United States (20):
  - Central Alabama Research, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of California Irvine, Orange, California
  - Johns Hopkins University School of Medicine, Washington D.C., District of Columbia
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Lakes Research LLC, Miami Lakes, Florida
  - Northwest Georgia Oncology Centers PC, Marietta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Revive Research Institute, Farmington Hills, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Revive Research Institute, Sterling Heights, Michigan
  - Upstate University Hospital, Syracuse, New York
  - White Plains Hospital Center for Cancer Care, White Plains, New York
  - Moses H Cone Memorial Hospital, Greensboro, North Carolina
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Lancaster General Hospital Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Kelsey Research Foundation, Houston, Texas
  - Best Cancer Care & Hematology, Houston, Texas
  - Lumi Research, Kingwood, Texas
- Australia (4):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - GenesisCare -North Shore (Oncology), St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
- France (4):
  - Centre Hospitalier Universitaire de Lyon - Hopital Edouard Herriot, Lyon Cédex 3
  - Institut regional du Cancer Montpellier, Montpellier
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Haut -lévêque, Pessac
- Germany (5):
  - Charite Universitaetsmedizin Berlin, Charité Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Carl Gustav Carus an der Technischen Universitaet Dresden, Dresden
  - Universitaetsmedizin Goettingen - Georg-August-Universitaet, Göttingen
  - Klinikum der Universitaet Muenchen Campus Grosshadern, München
  - Universitaetsklinikum der Eberhard Karls Universitaet Tuebingen, Tübingen
- Greece (7):
  - General Hospital of Athens Laiko, Athens
  - Evgenidio Hospital I Agia Trias, Athens
  - Hygeia Hospital, Athens
  - University Hospital of Heraklion, Heraklion - Crete
  - University Hospital of Patras, Pátrai
  - Theagenion Anticancer Hospital, Thessaloniki
  - Agios Loukas Clinic, Thessaloniki
- Italy (22):
  - Istituto Ospedaliero Fondazione Poliambulanza, Brescia
  - Azienda Ospedaliera Rilievo Nazionale e Alta Specializzazione Garibaldi Nesima, Catania
  - Azienda Ospedaliera Santa Croce e Carle, Confreria (CN)
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Azienda Sanitaria Locale 5 Spezzino Ospedale S Andrea, La Spezia
  - Azienda Unita Sanitaria Locale LE Presidio Ospedaliero Vito Fazzi Polo Oncologico Giovanni Paolo II, Lecce
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria di Cagliari Policlinico Duilio Casula, Monserrato CA
  - Azienda Ospedaliero Universitaria Luigi Vanvitelli, Napoli
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione Giovanni Pascale, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carita, Novara
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera Universitaria Pisana Ospedale Santa Chiara, Pisa
  - Azienda Ospedaliera San Carlo, Potenza
  - Azienda Unita Sanitaria Locale di Reggio Emilia Arcispedale Santa Maria Nuova, Reggio Emilia
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera San Giovanni Addolorata, Roma
  - Fondazione Policlinico Tor Vergata, Roma (RM)
  - Azienda Ospedaliera Cardinale Giovanni Panico, Tricase
  - Azienda Unita Locale Socio Sanitaria Berica 8, Vicenza
- Japan (15):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - St Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Hospital Organization Osaka National Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Mexico (3):
  - Health Pharma Professional Research SA de CV, Mexico City, Mexico City
  - Superare Centro de Infusion SA de CV, Mexico City, Mexico City
  - Trials In Medicine SC, Mexico City
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (10):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Complexo Hospitalario Universitario de Ourense, Ourense, Galicia
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital General Universitario de Elche, Elche, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario La Paz, Madrid
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- United Kingdom (6):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Free Hospital, London
  - Royal Marsden Hospital, London
  - Maidstone Hospital, Maidstone
  - Mount Vernon Cancer Centre, Northwood
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Fakih MG, Salvatore L, Esaki T, Modest DP, Lopez-Bravo DP, Taieb J, Karamouzis MV, Ruiz-Garcia E, Kim TW, Kuboki Y, Meriggi F, Cunningham D, Yeh KH, Chan E, Chao J, Saportas Y, Tran Q, Cremolini C, Pietrantonio F. Sotorasib plus Panitumumab in Refractory Colorectal Cancer with Mutated KRAS G12C. N Engl J Med. 2023 Dec 7;389(23):2125-2139. doi: 10.1056/NEJMoa2308795. Epub 2023 Oct 22. PMID 37870968
- [Background] Pietrantonio F, Salvatore L, Esaki T, Modest DP, Lopez-Bravo DP, Taieb J, Karamouzis MV, Ruiz-Garcia E, Kim TW, Kuboki Y, Meriggi F, Cunningham D, Yeh KH, Chan E, Chao J, Tran Q, Cremolini C, Fakih M. Overall Survival Analysis of the Phase III CodeBreaK 300 Study of Sotorasib Plus Panitumumab Versus Investigator's Choice in Chemorefractory KRAS G12C Colorectal Cancer. J Clin Oncol. 2025 Jul;43(19):2147-2154. doi: 10.1200/JCO-24-02026. Epub 2025 Apr 11. PMID 40215429
- [Background] Modest DP, Fakih M, Salvatore L, Esaki T, Lopez-Bravo DP, Taieb J, Karamouzis M, Ruiz-Garcia E, Kim TW, Kuboki Y, Meriggi F, Cunningham D, Yeh KH, Cremolini C, Tran Q, Chan E, Chao J, Majer IM, Pietrantonio F. Health-related quality of life in patients with KRASG12C-mutated chemorefractory metastatic colorectal cancer treated with sotorasib plus panitumumab or standard of care (CodeBreaK 300): results from a phase 3, randomised clinical trial. Lancet Oncol. 2025 Sep;26(9):1240-1251. doi: 10.1016/S1470-2045(25)00352-3. Epub 2025 Aug 11. PMID 40812325
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com